CLINICAL TRIAL: NCT06051240
Title: Lithium Treatment to Prevent Cognitive Impairment After Brain Radiotherapy
Acronym: LiBRA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-504071-24-00; 2023-504071-24-00 (Other: EudraCT)
Record Dates: First submitted 2023-06-12; First posted 2023-09-22 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-06

CONDITIONS: Cognitive Impairment; Cognitive Decline; Radiotherapy Side Effect; Radiotherapy; Complications; Brain Tumor; Memory Impairment; Late Effect of Radiation
Keywords: lithium; neuroprotection; neuroprotective; regenerative; prevention; radiation; pediatric brain tumor; brain tumor; cognition; cognitive
MeSH Terms: conditions — Cognitive Dysfunction; Radiation Injuries; Brain Neoplasms; Memory Disorders | interventions — Lithium; lithium sulfate

STUDY DESIGN:
Intervention Model Description: Randomization is based on whether or not the study participant had received radiotherapy to the whole brain (CSI) or only part of it (focal irradiation). Within each of these two arms there is a predetermined block randomization with a 2:1 lithium:placebo ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical-looking placebo is used. S-lithium levels are masked by using a separate lab service and sham values for placebo group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lithium (Experimental): Lithionit 42 mg (lithium sulphate, 6 mmol), start dose 1x1, then slow dose escalation using therapeutic drug monitoring (TDI) to establish a target serum level of 0.5-1.0 mmol/liter.
  Interventions: Drug: Lithium
- Placebo (Placebo Comparator): Identical looking placebo (white round tablet, 10 mm diameter) will be dose escalated and monitored the same way as lithium, with sham values guiding the dosing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium — Lithium sulphate, 42 mg (6 mmol lithium)
  Other Names: Lithionit; Lithium sulphate
  Arms: Lithium
Drug: Placebo — White round tablet, 10 mm. Identical to experimental drug (lithium)
  Arms: Placebo

SUMMARY:
Randomized, placebo-controlled, double-blinded, parallel group clinical trial to investigate if 6 months of oral lithium tablets (S-lithium 0,5-1,0 mmol/l) will prevent cognitive decline after brain radiotherapy in pediatric brain tumor survivors.

Primary outcome measure is Processing Speed Index (PSI) 2 years after start of study treatment.

DETAILED DESCRIPTION:
Late-appearing cognitive side effects after brain radiotherapy is a potential disabling condition in pediatric brain tumor survivors. It can have profound negative effects on education, career options and quality of life. There is no current interventional drug treatment to prevent this intellectual impairment after brain tumor treatment.

Primary objective:

To assess the efficacy of lithium treatment (up to 7 years) after brain radiotherapy (both whole brain and focal) for central nervous system malignancy in preventing late-appearing cognitive processing speed impairment in children aged 5 or older.

Secondary objectives:

* To assess the efficacy of lithium treatment through evaluation of other neuropsychological/quality of life test scores.
* To assess the efficacy of lithium treatment through evaluation of radiological findings after lithium treatment using Magnetic Resonance Imaging (MRI) of the brain.

Exploratory objectives:

To explore the feasibility, safety and tolerability of lithium treatment in this patient group, using side effect forms/adverse events (AE) reporting and laboratory measures.

ELIGIBILITY:
Inclusion Criteria:

* Age >5 years.
* Age <18 years at time of radiotherapy.
* Has received cranial/craniospinal radiation treatment of brain tumor within the last 7 years.
* Adequate contraceptive method to prevent pregnancy* during the entire lithium treatment period and six months thereafter.
* Negative pregnancy test* at screening, at start of study treatment, and monthly thereafter.
* Written informed consent from patient and/or caregiver.

Exclusion Criteria:

* Allergy/hypersensitivity to lithium or any of the excipients
* Renal failure (Cystatin C derived Glomerular Filtration Rate < 60).
* Cardiac failure or heart disease, including Brugada syndrome (or family history thereof).
* Uncontrolled hypothyroidism.
* Pregnancy or breast feeding.
* Severe fluid or electrolyte imbalance.
* Karnofsky-Lansky score < 60.
* Other condition deemed incompatible with inclusion in this study (estimated 2 year survival prognosis less than 25 %, expected poor protocol compliance, inability to swallow tablets, language difficulties).
* Inclusion in other study protocol precluding inclusion in this study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2033-08-31 (Estimated)

PRIMARY OUTCOMES:
Processing Speed Index (PSI) | 2 years after start of study treatment
  Cognitive processing speed. Normed score min 45, max 155. Higher = better.

SECONDARY OUTCOMES:
Fractional anisotropy (FA) index | Baseline (before treatment) - 5 years after start of study treatment
  White matter integrity on MRI brain.
Other Wechsler Intelligence scale scores (except PSI): | Baseline (before treatment) - 5 years after start of study treatment
  * Verbal Comprehension Index (VCI)
  * Visual Spatial Index (VSI)
  * Fluid Reasoning Index (FRI)
  * Working Memory Index (WMI)
  Normed score min 45, max 155. Higher = better.
Grooved pegboard | Baseline (before treatment) - 5 years after start of study treatment
  Motor speed / manual dexterity. Unit: time in seconds to complete all pegs. Lower=better.
Beery/Buktenica visual motor integration (VMI) | Baseline (before treatment) - 5 years after start of study treatment
  Visual motor integration. Normed score min 1, max 19. Higher = better.
Conner´s Continous Performance Test (CPT) III | Baseline (before treatment) - 5 years after start of study treatment
  Sustained attention. Multiple T-scores, min 0, max 80. Higher = better.
Delis-Kaplan Executive Function System Trail Making Test (D-KEFS TMT) | Baseline (before treatment) - 5 years after start of study treatment
  Executive function and inhibition, age 8 years and above. Normed score min 1, max 19. Higher = better.
Delis-Kaplan Executive Function System Color-Word Interference Test (D-KEFS CWT), age 8 years and above. | Baseline (before treatment) - 5 years after start of study treatment
  Executive function and inhibition. Normed score min 1, max 19. Higher = better.
Nepsy II: Inhibition, Verbal Fluency, | Baseline (before treatment) - 5 years after start of study treatment
  Executive function and inhibition, age below 8 years. Normed score min 1, max 19. Higher = better.
Pediatric QoL Inventory (PedsQL) | Baseline (before treatment) - 5 years after start of study treatment
  Health related quality of life. Score min 0, max 100. Higher=better.
University of California Los Angeles (UCLA) 3-Item Loneliness Scale (ULS-3) | Baseline (before treatment) - 5 years after start of study treatment
  Loneliness scale. Score min 3, max 9. Lower = better.
Strengths and Difficulties Questionnaire (SDQ) | Baseline (before treatment) - 5 years after start of study treatment
  Psychosocial strengths and difficulties. Score min 0, max 40.
Behavior Rating Inventory of Executive Function (BRIEF). | Baseline (before treatment) - 5 years after start of study treatment
  Executive function. Score min 20, max 80.

OTHER OUTCOMES:
Feasibility of recruitment and retention, numerical data | From screening - end of study (5 years)
  * Number of potentially eligible patients identified
  * Number of patients screened
  * Number of patients randomized
  * Number of patients completing the study per protocol
  * Number of patients terminating study during IMP treatment period (6 months).
  * Number of patients terminating study during follow-up period (up 5 years post IMP treatment)
Feasibility of recruitment and retention, qualitative data | From screening - end of study (5 years)
  * Description of reason why eligle patient declined screening
  * Description of reason why screened patient was not randomized/included
  * Description of reason(s) for early study termination.
Feasibility of treatment - IMP treatment duration | During study treatment (appx 6 months)
  Duration of IMP treatment, measured in total number of days where IMP was taken
Feasibility of treatment - number of IMP reductions and stops | During study treatment (appx 6 months)
  * Numbers of IMP dose reductions
  * Number of IMP temporary stops
Feasibility of treatment - reasons for IMP reductions and stops | During study treatment (appx 6 months)
  * Descriptions of reason(s) for IMP dose reductions
  * Descriptions of reason(s) for IMP temporary stops
  * Descriptions of reason(s) for IMP premature (before per protocol) permanent stop.
Feasibility of treatment - lithium serum concentration within target range | During study treatment (appx 6 months)
  * Number of target serum concentration measurements within target range (0.5-1.0 mmol/liter) divided by total number of measurements.
  * Number of target serum concentration measurements above target range (0.5-1.0 mmol/liter) divided by total number of measurments
  * Number of target serum concentration measurements below target range (0.5-1.0 mmol/liter) divided by total number of measurments
Feasibility of treatment - adverse events | During study treatment (appx 6 months) + 1 month
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Karolinska Universitetssjukhuset, Solna, Stockholm County
  - HOPE, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided